CLINICAL TRIAL: NCT06154356
Title: Effect of Action Observation and Motor Imagery Therapy on Balance, Functional Status and Quality of Life in Parkinson's Disease, Randomized Controlled Trial
Brief Title: Action Observation and Motor Imagery Therapy in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yurdagül Bahran Muştu, M.D., Principal investigator, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-2023/03
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation and motor imagery therapy for rehabilitation (Experimental): Action observation and motor imagery therapy for rehabilitation in Parkinson's Disease in addition to conventional rehabilitation programs.
  Interventions: Other: Action observation and motor imagery therapy for rehabilitation
- Sham action observation and motor imagery therapy for rehabilitation (Sham Comparator): Sham comparator for action observation and motor imagery therapy for rehabilitation in Parkinson's Disease in addition to conventional rehabilitation programs.
  Interventions: Other: Sham action observation and motor imagery therapy for rehabilitation

INTERVENTIONS:
Other: Action observation and motor imagery therapy for rehabilitation — Action observation; Patients will watch some exercises accompanied by music from a previously prepared video for 10 minutes. Exercises include 8-10 repetitions of abduction-adduction, horizontal abduction-adduction, flexion-extension and supination-pronation movements for the upper extremity, and stepping, forward-backward stepping, side stepping and ankle dorsiflexion movements for the lower extremity.
  Motor imagery training; Patients will be asked to visualize the actions they watched in their minds for 10 minutes.
  Then the patients will watch the video again and will be asked to perform the exercises while watching.
  Arms: Action observation and motor imagery therapy for rehabilitation
Other: Sham action observation and motor imagery therapy for rehabilitation — Sham action observation; Patients will watch a video consisting of static nature photographs for 10 minutes with the same music.
  Sham motor imaginary; Patients will think about the video they watched for 10 minutes.
  Then, they will watch another video in which the exercises are performed only once, and they will be asked to do the exercises. They will be given enough time to do 8-10 repetitions.
  Arms: Sham action observation and motor imagery therapy for rehabilitation

SUMMARY:
In recent years, motor imagery (MI) and action observation (AO) therapy strategies have been used in rehabilitation programs to increase motor learning in Parkinson's disease (PD). Visuomotor training strategies such as AO and MI therapy rely on the activity of the mirror neuron system to facilitate motor re-learning. Mirror neurons are activated during the performance of goal-directed actions, also when observing the same action and visualizing the action in the mind.

The aim of this clinical trial is to test whether the application of AO and MI treatment in PD in addition to conventional rehabilitation programs has an additional effect on Balance, Functional Status and Quality of Life.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disease with a chronic and progressive course. Freezing phenomena, gait disorders, and balance problems are common in PD. Gait and balance disorders and motor freezing attacks that occur as a result of PD increase the risk of falling, leading to a decrease in functional independence and quality of life. The main goal of Parkinson's rehabilitation is to ensure the maximum functional status and independence in daily living activities and to increase their quality of life.

In recent years, motor imagery (MI) and action observation (AO) therapy strategies have been used in rehabilitation programs to increase motor learning in PD. Visuomotor training strategies such as AO and MI therapy rely on the activity of the mirror neuron system to facilitate motor re-learning. Mirror neurons are activated during the performance of goal-directed actions, also when observing the same action and visualizing the action in the mind.

The aim of this clinical trial is to test whether the application of AO and MI treatment in PD in addition to conventional rehabilitation programs has an additional effect on Balance, Functional Status and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Parkinson's Disease
* Hoehn and Yahr Stage 1-3

Exclusion Criteria:

* Patients with cognitive dysfunction (those who cannot follow simple verbal instructions)
* Patients with severe hearing problems
* Patients with severe vision problems
* Patients with additional musculoskeletal system pathology that will affect physical performance (such as amputation, severe joint mobility limitation, peripheral nerve damage)
* Patients with uncontrolled hypertension and diabetes mellitus
* Patients with a history of symptomatic lung disease (such as asthma, chronic obstructive pulmonary disease, emphysema)
* Patients with a history of symptomatic cardiac disease (such as coronary artery disease, arrhythmia, heart failure)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The difference in the scores of the Berg Balance Scale between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Berg Balance Scale between pre- and post-rehabilitation assessments.
  Berg Balance Scale consists of 14 items. Total score ranges from 0 to 56. Higher scores indicate better balance.
The difference in the scores of the The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale between pre- and post-rehabilitation assessments.
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) consists of four sections: Part 1: non-motor experiences of daily living, Part 2: motor experiences of daily living, Part 3: motor examination, Part 4: motor complications. It consists of a total of 50 questions. In this study, sections II (motor experiences of daily living) and III (motor examination) will be used. Each item is is scored between 0 and 4. Higher values indicate that the patient's condition is worse.
The difference in the scores of the Timed Up and Go Test between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Timed Up and Go Test between pre- and post-rehabilitation assessments
The difference in the scores of the Five Times Sit to Stand Test between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Five Times Sit to Stand Test between pre- and post-rehabilitation assessments

SECONDARY OUTCOMES:
The difference in the scores of the Parkinson's Disease Questionnaire between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Parkinson's Disease Questionnaire (PDQ-39) between pre- and post-rehabilitation assessments.
  Parkinson's Disease Questionnaire consists of a total of 39 items and eight subgroups. In the survey, each item is scored between 0 and 4. Lower scores indicate better quality of life.
The difference in the scores of the Freezing of Gait Questionnaire between pre- and post-rehabilitation assessments | 6 weeks
  Univariate statistical analyses will be performed to calculate differences in the scores of the Freezing of Gait Questionnaire between pre- and post-rehabilitation assessments.
  Freezing of Gait Questionnaire consists of six questions. Each question has a 5-point scale, where 0 means an absence of symptoms and 4 represents the worst stage. The total score on the Freezing of Gait Questionnaire ranges from 0 to 24 points. The higher the score is, the more the Freezing of Gait is pronounced.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagul Bahran Mustu, MD., Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Karaman, Turkey (Türkiye)